CLINICAL TRIAL: NCT05311176
Title: nextHERIZON: An Open-Label, Signal Generating, Phase 2 Study of HER-Vaxx in Combination With Chemotherapy or Pembrolizumab in Patients With Metastatic HER2/Neu Over-Expressing Gastric or Gastroesophageal Junction (GEJ) Adenocarcinomas Who Have Previously Received Trastuzumab and Progressed on This Treatment
Brief Title: A Study of IMU-131 (HER-Vaxx) in Combination With Chemotherapy or Pembrolizumab in Patients With Metastatic HER2/Neu Over-Expressing Gastric Cancer (nextHERIZON)
Acronym: nextHERIZON
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was discontinued because of slow enrollment and organizational priorities and not because of any findings related to safety or efficacy.
Sponsor: Imugene Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMU.131.203
Record Dates: First submitted 2022-03-08; First posted 2022-04-05 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer; Cancer of Stomach; Gastric Adenocarcinoma; Stomach Cancer; Stomach Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: HER2; Immunotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Ramucirumab; Paclitaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: HER-Vaxx in combination with chemotherapy (ramucirumab plus paclitaxel) (Experimental): Patients who have received an immune checkpoint inhibitor (ICI) previously will exclusively be enrolled in Arm 1 treated with HER-Vaxx (IM) in combination with chemotherapy (ramucirumab plus paclitaxel)
  Interventions: Biological: IMU-131; Drug: Ramucirumab plus Paclitaxel
- Arm 2: HER-Vaxx in combination with pembrolizumab (Experimental): Arm 2 will investigate the combination of HER-Vaxx plus pembrolizumab in patients who are naïve to ICI treatment including patients who have had chemotherapy only treatment after progression on trastuzumab. As the combination treatment has not been investigated, Arm 2 is planned to initiate with a safety run-in phase.
  Interventions: Biological: IMU-131; Biological: Pembrolizumab

INTERVENTIONS:
Biological: IMU-131 — IMU-131 will be administered intramuscularly into the deltoid region of the arm on Day 1, 15, 29 and 57 and then every 63 days until disease progression or treatment discontinuation.
  Other Names: HER-Vaxx
Drug: Ramucirumab plus Paclitaxel — Chemotherapy to be administered every 3 weeks (Q3W) starting on Day 1.
  Other Names: Standard of Care Chemotherapy
  Arms: Arm 1: HER-Vaxx in combination with chemotherapy (ramucirumab plus paclitaxel)
Biological: Pembrolizumab — Pembrolizumab will be administered every 3 weeks (Q3W) starting on Day 1 until disease progression or treatment discontinuation.
  Other Names: Keytruda
  Arms: Arm 2: HER-Vaxx in combination with pembrolizumab

SUMMARY:
This is a Phase 2, signal generating, open-label, 2-Arm, non-randomized study, in patients with metastatic HER2/neu over-expressing gastric cancer or gastroesophageal adenocarcinomas.

DETAILED DESCRIPTION:
It is hypothesized that the introduction of HER-Vaxx after 1L treatment in patients that have progressed under trastuzumab may overcome potential resistance against trastuzumab in combination with chemotherapy and can be continued after chemotherapy is terminated. Based on pre-clinical data HER-Vaxx may also synergize with pembrolizumab and therefore serve as a potentially better tolerated and chemotherapy-free treatment opportunity in metastatic patients that progressed under their previous therapy.

The study is designed to generate safety data and efficacy signals to support further development of HER-Vaxx in ≥2L mGC/GEJ cancer after progression with trastuzumab.

The study includes two treatment arms that will be analyzed independently using a 2-Stage design:

* Arm 1: HER-Vaxx in combination with chemotherapy (ramucirumab plus paclitaxel)
* Arm 2: HER-Vaxx in combination with pembrolizumab.

All patients must have received trastuzumab and progressed after 1L to be eligible for enrolment. Patients who have received an immune checkpoint inhibitor (ICI) previously will exclusively be enrolled in Arm 1 (HER-Vaxx + chemotherapy). Patients who are naïve to ICI treatment will exclusively be enrolled into Arm 2 (HER-Vaxx + pembrolizumab).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years with confirmed diagnosis of advanced or metastatic HER2/neu overexpressing gastric or GEJ adenocarcinoma;
2. Progressed on or after trastuzumab therapy;
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
4. Life expectancy of a minimum of 3 months;
5. At least one measurable lesion as defined by RECIST 1.1 criteria and assessed by the local investigator;
6. HER2/neu overexpression assessed using post-progression fresh or archival tissue, or post-progression pathology report;
7. Adequate left ventricular ejection function at baseline, defined as left ventricular ejection fraction (LVEF) > 50% by echocardiogram or Multi Gated Acquisition (MUGA) scan;
8. Adequate hematologic, liver and renal function;
9. A female patient of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 120 days after the last dose of assigned treatment.

Exclusion Criteria:

1. Previous malignant disease (other than primary malignancy) within the last 5 years, except basal or squamous cell carcinoma of the skin or cervical carcinoma in situ;
2. Concurrent active malignancy except for adequately controlled limited basal cell carcinoma of the skin;
3. Systemic chemotherapy or major surgery within 28 days before starting study treatment and recovered from all adverse events ≤ Grade 1 or baseline with possible exceptions for neuropathy and endocrine-related AEs;
4. Received prior radiotherapy within 2 weeks of start of study treatment and recovered from all radiation-related toxicities and not require corticosteroids; or history of radiation pneumonitis.
5. Previous treatment with trastuzumab-deruxtecan or any other anti-HER2 therapy (except trastuzumab);
6. Clinically significant cardiovascular disease, or other diseases that in the Investigator's opinion may influence the patient's tolerance to study treatment;
7. Pleural effusion or ascites requiring more than weekly drainage;
8. Prior organ transplantation, including allogenic stem-cell transplantation;
9. Chronic immunosuppressive therapy within 7 days prior the first dose of study drug;
10. Active, known, or suspected autoimmune disease;
11. History of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease;
12. Positivity for human immunodeficiency virus (HIV) (HIV 1/2 antibodies) or active hepatitis B (HBsAg reactive) or active hepatitis C (HCV ribonucleic acid [RNA] qualitative) infection;
13. Current participation or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment;
14. Any vaccination within 30 days prior to starting study treatment;
15. Pregnant or lactating females;
16. Arm 2 only: Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent;
17. Arm 2 only: Has received prior therapy with an ICI or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) and was discontinued from treatment due to a grade 3 or higher adverse event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (2):
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - The Queen Elizabeth Hospital, Woodville South, South Australia
- Taiwan (5):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Imugene Limited — http://www.imugene.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 7 participants were enrolled in the trial. A second arm was planned with IMU 131 + chemotherapy (ramucirumab and paclitaxel) but did not enroll any participants.
Groups:
- IMU-131 + Pembrolizumab: Participants received IMU-131 intramuscularly (IM) on Day 1, 15, 29 and 57 and then every 63 days until disease progression or treatment discontinuation. Pembrolizumab was administered every 3 weeks (Q3W) starting on Day 1 until disease progression or treatment discontinuation.
Period: Overall Study
Arm/Group | IMU-131 + Pembrolizumab
Started | 7
Received at Least 1 Dose of Study Drug | 7
Completed | 0
Not Completed | 7
Not completed — Death | 6
Not completed — Sponsor discontinued the study | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAF) included all participants who received at least 1 dose of study treatment.
Groups:
- IMU-131 + Pembrolizumab: Participants received IMU-131 IM on Day 1, 15, 29 and 57 and then every 63 days until disease progression or treatment discontinuation. Pembrolizumab was administered Q3W starting on Day 1 until disease progression or treatment discontinuation.
Arm/Group | IMU-131 + Pembrolizumab
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (6.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in the Reported AE section.
Time Frame: First dose of study drug up to approximately 1.5 years
Population: The Safety Analysis Set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-131 + Pembrolizumab
Number analyzed (Participants) | 7
Participants | 6

2. Primary Outcome: Number of Participants With Immune-related Adverse Events (irAEs)
Description: irAEs were monitored throughout the study as per National Comprehensive Cancer Network® (NCCN) guidelines. irAEs were defined as any Grade ≥3 event that did not resolve to Grade 1 (or baseline) within 7 days from the onset of the event, or any Grade ≥3 organ toxicity involving major organ systems that persisted for greater than 72 hours.
Time Frame: First dose of study drug up to approximately 1.5 years
Population: The Safety Analysis Set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-131 + Pembrolizumab
Number analyzed (Participants) | 7
Participants | 1

3. Primary Outcome: Number of Participants With Objective Response
Description: Objective response was defined as the number of participants achieving a confirmed best overall response of complete response (CR) or partial response (PR) according to Response Evaluation Criteria for Solid Tumors, Version 1.1 (RECIST v1.1).
  * CR: Disappearance of all target lesions.
  * PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to approximately 6 months
Population: The evaluable analysis set included all participants who received at least 1 administration of study treatment and had an evaluable baseline tumor assessment and had at least one evaluable post-baseline tumor response assessment as per RECIST v1.1, or were discontinued due to toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-131 + Pembrolizumab
Number analyzed (Participants) | 5
Participants | 0

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from first dose of study drug to death due from any cause.
Time Frame: Up to approximately 6 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMU-131 + Pembrolizumab
Number analyzed (Participants) | 5
months | NA [NA to NA] — OS could not be calculated due to insufficient number of events.

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from first dose of study drug to first documentation of progressive disease (PD) based on RECIST 1.1, or to death from any cause.
  PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: Up to approximately 6 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMU-131 + Pembrolizumab
Number analyzed (Participants) | 5
months | NA [NA to NA] — PFS could not be calculated due to insufficient number of events.

6. Secondary Outcome: Duration of Response (DoR)
Description: DoR was measured from earliest CR or PR until first documentation of PD based on RECIST 1.1 or death due to any cause.
Time Frame: Up to approximately 6 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMU-131 + Pembrolizumab
Number analyzed (Participants) | 5
months | NA [NA to NA] — DoR could not be calculated due to insufficient number of events.

ADVERSE EVENTS:
Time Frame: First dose of study drug up to approximately 1.5 years
Groups:
- IMU-131 + Pembrolizumab: Participants received IMU-131 IM on Days 1, 15, 29 and 57 and then every 63 days until disease progression or treatment discontinuation. Pembrolizumab was administered Q3W starting on Day 1 until disease progression or treatment discontinuation.
Arm/Group | IMU-131 + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 6/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMU-131 + Pembrolizumab (N=7)
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Pain (General disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Oral candidiasis (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Brain oedema (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Speech disorder developmental (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Some efficacy endpoints could not be analyzed because the study was discontinued after only a small number of participants had been enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT05311176/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT05311176/SAP_001.pdf